CLINICAL TRIAL: NCT02100163
Title: Controling Pain After Orthopedic Trauma
Brief Title: Virtual Reality Pain Control Orthopedic Trauma
Acronym: VROT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, David R. Patterson, Professor, National Institute of General Medical Sciences (NIGMS)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 43654-J/001500
Record Dates: First submitted 2014-03-19; First posted 2014-03-31 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Trauma/Injury Problem
Keywords: Ortho trauma. Virtual Reality. Pain. Anxiety
MeSH Terms: conditions — Accidental Injuries

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Virtual Reality Hypnosis (Experimental): The patient receives VRH daily.
  Interventions: Behavioral: Virtual Reality Hypnosis
- Audio Hypnosis (Experimental): The patient receives Audio Hypnosis daily.
  Interventions: Behavioral: Audio Hypnosis
- Standard Treatment (Experimental): The patient receives the standard treatment. This is a control group and there are no interventions.
  Interventions: Other: Standard treatment

INTERVENTIONS:
Behavioral: Virtual Reality Hypnosis — The patient receives virtual reality hypnosis daily.
  Other Names: VRH
  Arms: Virtual Reality Hypnosis
Behavioral: Audio Hypnosis — Patient will listen to an Audio Hypnosis recording daily.
  Arms: Audio Hypnosis
Other: Standard treatment
  Other Names: Tere are no interventions
  Arms: Standard Treatment

SUMMARY:
The treatment of postoperative pain after severe trauma is poorly understood, and it can lead to chronic pain, opiate drug addiction and elevated health care costs. The proposed project will be a randomized controlled trial to evaluate an innovative methodology for delivering clinical hypnosis (virtual reality hypnosis) for pain control as well as a more time-honored delivery system that uses audio recordings. The goal will be to reduce postoperative pain in a sample of patients hospitalized for the care of severe orthopedic trauma and other types trauma. This proposal will test innovative and low-risk approaches to reducing postoperative trauma pain that are designed to reduce pain, anxiety and other complications after surgery. The findings have the potential not only to reduce pain and suffering in patients who have suffered severe trauma but could be applicable to the millions of people who have surgery every year. Reducing addictive opiate-based medication and health care costs are both potential outcomes from this project.

ELIGIBILITY:
Inclusion Criteria:

* Compliant and able to complete questionnaires
* English speaking
* Hospitalization for trauma orthopedic injuries
* No history of psychiatric disorder
* Not demonstrating delirium, psychosis or any form of Organic Brain Disorder
* Able to communicate verbally
* 18 years of age or older

Exclusion Criteria:

* Not capable of filling out study measures
* Evidence of a traumatic brain injury or any other
* Cognitive deficits that would impact decisional capacity to consent for the
* study or complete measures
* History of psychiatric disorder as evidenced in the RN and MD admission notes
* Unable to communicate verbally
* Extreme susceptibility to motion sickness
* Seizure history
* Non-English speaking
* In isolation for infections such as Clostridium difficile

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2018-06-24 (Actual); Study Completion 2018-06-24 (Actual)

PRIMARY OUTCOMES:
Graphic Rating Scale (GRS) pain and anxiety Questionnaire | up to 10 days
  Measures pain and anxiety

SECONDARY OUTCOMES:
Tellegen Absorption Scale | 1 day (Once in the hospital)
  consists of 34 true-false items that examines hypnotic susceptibility in individuals

OTHER OUTCOMES:
The Short Stanford Hypnotizability Scale (SSHS) | 1 day (Once in the hospital)
  assesses hypnotizability with five items: moving hands together motor suggestion, a dream within hypnosis, age regression, a posthypnotic suggestion of a cough, and posthypnotic amnesia.
SF-36 | 1 day (Once in the hospital)
  self-reported survey to measure health status and quality of life
Brief Symptom Inventory | 1 day (Once in the hospital)
  self-reported instrument that measures the current overview of psychological symptoms and their intensity

CONTACTS AND LOCATIONS:
Overall Officials: David R. Patterson, Ph.D., Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States